CLINICAL TRIAL: NCT00037648
Title: A Randomized, Multi-center, Blinded, Placebo-controlled Study With an Open-label Run-in Period to Evaluate the Efficacy, Safety, and Pharmacokinetics of Daily, Single, Subcutaneous Injections of r-metHuIL-1ra (Anakinra) in Polyarticular-Course Juvenile Rheumatoid Arthritis
Brief Title: Juvenile Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Organization: Swedish Orphan Biovitrum (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 990758-990779
Record Dates: First submitted 2002-05-17; First posted 2002-05-20 (Estimated); Last update posted 2009-11-26 (Estimated); Status verified 2008-02

CONDITIONS: Juvenile Chronic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- anakinra (Experimental)
  Interventions: Drug: Anakinra

INTERVENTIONS:
Drug: Anakinra — anakinra
  Arms: anakinra
Drug: Placebo — placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to determine the safety of anakinra in patients with Polyarticular-Course Juvenile Rheumatoid Arthritis, a form of rheumatoid arthritis affecting children.

ELIGIBILITY:
* Male or female age 2-17 yrs inclusive * Minimum weight 10 KG * Diagnosis of Chronic Arthritis

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 86 (Actual)
Dates: Start 2000-07; Primary Completion 2003-11 (Actual); Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
The primary outcome of the study was to evaluate the safety of anakinra | 28 weeks

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com